CLINICAL TRIAL: NCT01937117
Title: A Phase 2 Clinical Trial Assessing the Correlation of Early Changes in Standardized Uptake Value (SUV) on Positron Emission Tomography (PET) With Pathological Complete Response (pCR) to Pertuzumab and Trastuzumab in Patients With Primary Operable HER2-Positive Breast Cancer
Brief Title: Pertuzumab and Trastuzumab as Neoadjuvant Treatment in Patients With HER2-Positive Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBCRC 026; TBCRC026 (Other: Translational Breast Cancer Research Consortium (TBCRC)); NA_00080994 (Other: JHMIRB)
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Preoperative treatment; Neoadjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trastuzumab and Pertuzumab (Experimental): Preoperative treatment with trastuzumab (8 mg/kg loading dose, then 6 mg/kg every 3 weeks, IV) and pertuzumab (840 mg as a loading dose, then 420 mg every 3 weeks, IV) every 3 weeks for 4 doses (total 12 weeks or 3 months of treatment) as assessed by Positron Emission Tomography (PET)
  Interventions: Procedure: Positron emission tomography (PET); Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Procedure: Positron emission tomography (PET) — PET will be performed at baseline and on day 15
  Other Names: FDG PET, PET/CT
Drug: Trastuzumab — 8 mg/kg loading dose, then 6 mg/kg every 3 weeks, IV
  Other Names: Herceptin
Drug: Pertuzumab — 840 mg as a loading dose, then 420 mg every 3 weeks, IV
  Other Names: Perjeta

SUMMARY:
This research is being done to determine if early changes on a type of imaging procedure called PET (Positron Emission Tomography) can predict which patients are most likely to respond to the combination of trastuzumab and pertuzumab when given prior to surgery.

DETAILED DESCRIPTION:
This study will evaluate for the first time the correlation between early changes in SUV and pCR in men and women with ER-negative, human epidermal growth factor receptor 2 (HER2)-positive breast cancer receiving trastuzumab and pertuzumab (PT) pre-operatively. This has not previously been evaluated in patients receiving anti HER2 therapy alone and as such is novel and potentially practice changing. The results from this phase 2 biomarker study will be used to plan a randomized study using a predefined cut point for SUV decline such that the investigators can further attempt to identify a group of individuals with HER2-positive early breast cancer who do not require cytotoxic chemotherapy in addition to anti-HER2 agents. This non-invasive biomarker approach will be of great interest to breast cancer oncologists and patients by facilitating a personalized approach to managing patients with HER2-positive disease that will undoubtedly spare toxicity and reduce the costs associated with anti-cancer strategies, without compromising efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, 18 years old or older
* Histologically proven infiltrating carcinoma of the breast on core needle biopsy that is: estrogen receptor (ER)/progesterone receptor (PR) ≤10% staining by immunohistochemistry (IHC) and HER2 positive - IHC 3+, in situ hybridization (ISH) ≥2.0, or average HER2 copy number ≥6.0 signals per cell or per current American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) or National Comprehensive Cancer Network (NCCN) guidelines. Note: All histological diagnostic material should be reviewed at enrolling institution as required per local standards.
* Unresected, untreated breast cancer that meets one of the following clinical stages (see Appendix A): T2, T3, or T4a-c lesion, any N, M0. Note: Patients with inflammatory breast cancer (T4d) are not eligible. Bilateral cancers are permitted with approval of the Protocol Chair.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Appendix B)
* Adequate organ function as follows:

  1. Absolute neutrophil count (ANC) ≥ 1,500/mm3
  2. Platelet count ≥ 100,000/mm3
  3. Hemoglobin ≥ 10 g/dL
  4. Creatinine ≤ 1.5 times the upper limit of normal with creatinine clearance ≥ 50 mL/min using the Modified Cockcroft-Gault method
  5. Bilirubin (total) ≤ 1.5 times upper limit normal (with exception of Gilberts syndrome)
  6. AST(SGOT), ALT(SGPT), and alkaline phosphatase ≤ 2 times the upper limit of normal
* Adequate cardiac function as defined by left ventricular ejection fraction (LVEF) ≥ 50% on echocardiogram or multi-gated acquisition scan (MUGA)
* Able and amenable to baseline and follow-up PET/CT imaging and study-specific biopsy procedures. Note: If there are any imaging concerns that the patient may not be suitable for quantitative PET/CT (e.g., a metallic device directly overlies the breast), discussion with the local and central radiologists is required to confirm eligibility for the trial. Also, it is expected that subjects have all PET/CT imaging done on pre-qualified machines for the study; if baseline imaging done on another machine, please contact the Protocol Chair/designee for guidance prior to confirming eligibility.
* The patient, if of childbearing potential, is willing to use effective, non-hormonal contraception while on treatment and for at least 6 months following the last dose of therapy.
* Patient understands the study regimen, its requirements, risks, and discomforts, and is able and willing to sign an informed consent form.

Exclusion Criteria:

* Received prior or ongoing local (e.g radiation) or systemic treatment (chemotherapy or endocrine therapy) for the current breast cancer. Patients who received tamoxifen or raloxifene or another agent for prevention of breast cancer may be included as long as the patient has discontinued the treatment at least one month prior to baseline study biopsy.
* Systemic treatment for prior cancer within the last 5 years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
* Women who are pregnant or nursing
* Current use of any investigational agents
* Known hypersensitivity to trastuzumab or pertuzumab
* Any medical condition that in the opinion of the investigator puts the patient at risk of potentially serious complications while on this therapy. Specifically, uncontrolled hypertension (systolic >150 and/or diastolic >100), unstable angina, congestive heart failure of any New York Heart Association (NYHA) classification, serious cardiac arrhythmia requiring treatment (exception: atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infarction within 6 months of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roisin Connolly, MBBCh, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (10):
- United States (10):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Johns Hopkins Kimmel Cancer Center at Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data.

REFERENCES:
- [Result] Connolly RM, Leal JP, Solnes L, Huang CY, Carpenter A, Gaffney K, Abramson V, Carey LA, Liu MC, Rimawi M, Specht J, Storniolo AM, Valero V, Vaklavas C, Krop IE, Winer EP, Camp M, Miller RS, Wolff AC, Cimino-Mathews A, Park BH, Wahl RL, Stearns V. TBCRC026: Phase II Trial Correlating Standardized Uptake Value With Pathologic Complete Response to Pertuzumab and Trastuzumab in Breast Cancer. J Clin Oncol. 2019 Mar 20;37(9):714-722. doi: 10.1200/JCO.2018.78.7986. Epub 2019 Feb 5. PMID 30721110 (Retraction: PMID 33999659 J Clin Oncol. 2021 Jul 10;39(20):2319)
- [Derived] Hennessy MA, Cimino-Mathews A, Carter JM, Kachergus JM, Ma Y, Leal JP, Solnes LB, Denbow R, Abramson VG, Carey LA, Rimawi M, Specht J, Storniolo AM, Valero V, Vaklavas C, Winer EP, Krop IE, Wolff AC, Wahl RL, Perez EA, Huang CY, Stearns V, Thompson EA, Connolly RM. Multiplex Spatial Proteomic Analysis of HER2-Positive Breast Tumors Reveals Unique Molecular and Immunologic Features Associated With Treatment Response. JCO Precis Oncol. 2025 Apr;9:e2400546. doi: 10.1200/PO-24-00546. Epub 2025 Apr 3. PMID 40179327

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trastuzumab and Pertuzumab
Started | 88
Completed | 75
Not Completed | 13
Not completed — Disease Progression | 7
Not completed — Physician Decision | 4
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab and Pertuzumab
Number analyzed (Participants) | 88
Age, Continuous [Median (Standard Deviation); unit: years] | 58 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 75
  Black or African American | 7
  Other | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale measures performance status, with scores ranging from 0-5; 0= fully active, performs without restriction, 1= can ambulate, but restricted in physically strenuous activity, 2= ambulatory and capable of self-care, but unable to work, active for >50% of waking hours, 3= limited self-care, confined to bed or chair for >50% of waking hours, 4= completely disabled, totally confined to bed/chair, 5= deceased
  Participants
    0 | 76
    1 | 12
Baseline clinical tumor size [Median (Standard Deviation); unit: cm] — Primary breast tumor size in centimeters (cm)
  cm | 3.7 (2)
Clinical tumor T staging [Count of Participants; unit: Participants] — T refers to the extent (size) of the tumor and is based off the staging system used for breast cancer is the American Joint Committee on Cancer (AJCC). Staging is as follows: T1= tumor <= 2cm in greatest dimension, T2= tumor >2cm in greatest dimension, T3= tumor >5cm in greatest dimension, and T4= tumor of any size with direct extension to chest wall (T4a) or skin (T4b). A higher number reflects a more progressive stage.
  Participants
    T1 | 0
    T2 | 66
    T3 | 19
    T4 | 3
Baseline clinical nodal status [Count of Participants; unit: Participants] — Based from the American Joint Committee on Cancer (AJCC) TNM system, this measures whether participants' cancer has spread to lymph nodes near the breast.
  Participants
    Negative | 45
    Positive | 43
Clinical tumor N staging [Count of Participants; unit: Participants] — AJCC staging: N0= no regional lymph node (LN) metastasis ("mets"), N1= mets in movable ipsilateral axillary LN; N2= mets in ipsilateral axillary LNs fixed or matted, or in clinically apparent ipsilateral internal mammary LN without of clinically evident axillary LN mets; N3= mets in ipsilateral infraclavicular LN, or in clinically apparent ipsilateral internal mammary LNs and in the presence of clinically evident axillary LN mets; or mets in ipsilateral supraclavicular LN with or without axillary or internal mammary lymph node involvement. A higher number reflects a greater region of mets.
  Participants
    N0 | 45
    N1 | 38
    N2 | 3
    N3 | 2
Baseline clinical stage [Count of Participants; unit: Participants] — Based on AJCC TNM staging (as described above): earliest stage breast cancers are stage 0 (carcinoma in situ). It then ranges from stage I (1) through IV (4), with a higher stage reflecting worse outcome. Stage I= T1N0M0, Stage II= T0N1M0, T1N1M0, T2N0M0, T2N1M0, T3N0M0, Stage III= T0N2M0, T1N2M0, T2N2M0, T3N1M0, T3N2M0, T4N0M0, T4N1M0, T4N2M0, any TN3M0.
  Participants
    Stage I | 0
    Stage II | 74
    Stage III | 14
    Stage IV | 0
Tumor Grade [Count of Participants; unit: Participants] — Tumor grade measures how much the cancer cells look like normal cells. Grading is as follows: Grade 1 (well differentiated)= the cells are slower-growing, and look more like normal breast tissue; Grade 2 (moderately differentiated)= the cells are growing at a speed of and look like cells somewhere between grades 1 and 3, Grade 3 (poorly differentiated) = the cells look very different from normal cells and will probably grow and spread faster. A higher grade reflects a worse prognosis.
  Participants
    Grade 1 | 0
    Grade 2 | 22
    Grade 3 | 66
Additional neoadjuvant therapy [Count of Participants; unit: Participants] — Study treatment was pertuzumab and trastuzumab. If required by care team, participants could receive additional treatment, outside of the protocol, prior to surgery.
  Participants
    Yes | 25
    No | 59
    N/A | 4
Type of Surgery [Count of Participants; unit: Participants] — Type of surgical intervention received.
  Participants
    Mastectomy | 51
    Breast-conserving therapy | 33
    N/A | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Standardized Uptake Value (SUV) as Measured by SULmax on [18F]Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)
Description: SULmax is the maximum SUV corrected for lean body mass. Change in SULmax from baseline to Day 15 on FDG PET in correlation with pathological complete response (pCR) in patients treated with preoperative pertuzumab/trastuzumab. pCR was defined as no viable invasive cancer in breast and axilla by local pathology review. SULmax was measured via spherical volume over the target primary breast cancer tissue.
Time Frame: Baseline and Day 15
Population: Data was evaluable in only 83/88 participants.
Measure: Mean (Standard Deviation); unit: percent reduction in SULmax
Arm/Group | Trastuzumab and Pertuzumab
Number analyzed (Participants) | 83
percent reduction in SULmax
  pCR: number analyzed (Participants) | 28
  pCR | 61.9 (22.3)
  no pCR: number analyzed (Participants) | 55
  no pCR | 34.3 (31.9)

2. Secondary Outcome: Change in ptDNA With Response
Description: To correlate PIK3CA mutation status and other genomic alterations (mutations/somatic rearrangements) qualitatively and quantitatively in plasma tumor DNA (ptDNA) with pCR
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2026-05

3. Secondary Outcome: Change in PI3K Pathway Activation With Response
Description: To correlate PI3K pathway activation (e.g. PTEN low and/or PIK3CA mutation, human epidermal growth factor receptor (HER) 1-4 expression and/or phosphorylation) in tumor samples and pCR
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: Changes in Ki67 With Response
Description: To correlate baseline and change (day 15) in Ki67 with pCR
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Trastuzumab and Pertuzumab
All-Cause Mortality (participants affected / at risk) | 0/88
Serious Adverse Events (participants affected / at risk) | 2/88
Other Adverse Events (participants affected / at risk) | 88/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab and Pertuzumab (N=88)
Sepsis (Injury, poisoning and procedural complications) | 1 (2) — Not related to study product.
Enterocolitis (Gastrointestinal disorders) | 1 (1) — Not related to study product.
OTHER ADVERSE EVENTS (reported when occurring in more than 4.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab and Pertuzumab (N=88)
Rash (NOS) (Skin and subcutaneous tissue disorders) | 17 (17)
Diarrhea (Gastrointestinal disorders) | 80 (80)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Mucositis (Gastrointestinal disorders) | 12 (12)
Nausea (Gastrointestinal disorders) | 24 (24)
Fatigue (General disorders) | 30 (30)
Headache (Nervous system disorders) | 13 (13)
Chills (General disorders) | 10 (10)
Dysgeusia (Nervous system disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT01937117/Prot_SAP_001.pdf